CLINICAL TRIAL: NCT07255144
Title: Ultrafast Ultrasound Imaging: Application in Pediatric Cardiology: Cardiac Ultrafast
Brief Title: Ultrafast Ultrasound Imaging in Pediatric Cardiology
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2024/52; CER-BDX 2024-169 (Other: Comité d'étique - Centre Ethique et Recherche en Santé de Bordeaux)
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: CHD - Congenital Heart Disease
Keywords: Congenital heart disease; Paediatric; Cardiac Imaging; Ultrafast ultrasounf
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CHD: Patients with CHD
  Interventions: Other: Cardiac Ultrafast Ultrasound
- General population: General population patients in good general health as evidenced by medical history coming to our department for a check-up OR diagnosed with small Atrial Septal Defect or small Patent Foramen Ovale
  Interventions: Other: Cardiac Ultrafast Ultrasound

INTERVENTIONS:
Other: Cardiac Ultrafast Ultrasound — Ultrafast ultrasound imaging(UFUS), ultrasound images at a very high rate, using a Verasonics system (ultrasound open platform).

SUMMARY:
About 13 in 1000 children are born with heart disease. Current tools poorly assess heart filling in children, limiting treatment. This study explores ultrafast ultrasound imaging to measure heart stiffness and perfusion in children with congenital heart disease.

DETAILED DESCRIPTION:
About 13/1000 children are born with heart disease. As a result of better treatment, there is an increasing population of children surviving with congenital heart disease (CHD) as well as a growing number of children with obesity, hypertension and serious chronic diseases, such as cancer and kidney disease, who are at risk of developing heart disease. All of these diseases affect the heart muscle and one of the main mechanisms resulting in heart muscle damage is the development of scar tissue (fibrosis). Fibrosis makes the heart muscle stiffer and therefore more difficult to fill. The heart must fill properly with blood in order to function well; but it is very difficult to study the filling of the heart using current diagnostic tools. One of the main challenges in pediatric cardiology is that non-invasive diagnostic approaches used in adult patients to assess heart filling (diastolic function) have proven inadequate in children. This knowledge gap has limited therapeutic progress in this vulnerable population; and to date there is no effective therapy that improves the filling of the heart.

The aim of this study is to explore new potential of ultrasound to assess diastolic function in CHD children. Ultrafast ultrasound imaging (UFUS), consisting of ultrasound images at a very high rate, is a new ultrasound approach to assess cardiac function.

Using a Verasonics system (ultrasound open platform), we will assess the myocardial stiffness and the myocardial perfusion by UFUS.

ELIGIBILITY:
Inclusion Criteria:

* Every patient of CHD department of any age or any sex:

  * Patients with CHD
  * General population patients in good general health as evidenced by medical history coming to our department for a check-up OR diagnosed with small Atrial Septal Defect or small Patent Foramen Ovale
* Social security affiliation
* Parental or legal guardian's non-opposition

Exclusion Criteria:

* Arrhythmia
* Segmental kinetic disorder.
* Pacemaker or multisite stimulation, defibrillator,
* Anechoic
* Allergy to echocardiography gel.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Every patient of CHD department of any age or any sex: 300 participants including 100 general population patients and 200 patients with CHD
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2028-03-11 (Estimated); Study Completion 2028-03-11 (Estimated)

PRIMARY OUTCOMES:
Myocardial stiffness | Baseline
  assessed with ultrasound data processed using the Verasonics system, to evaluate diastolic function
Myocardial perfusion | Baseline
  assessed with ultrasound data processed using the Verasonics system, to evaluate diastolic function

SECONDARY OUTCOMES:
Echocardiographic parameters | Baseline
  3. Echocardiographic parameters according to international guidelines for screening for structural or functional intra-cardiac abnormalities (Lopez et al. JASE. 2024) and assessed by conventional ultrasound and ultrafast ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Cardiologique Haut Lévêque, Pessac, France, France